CLINICAL TRIAL: NCT01734915
Title: Detecting EGFR T790M Mutations From Circulating Tumor Cells
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Memorial Sloan Kettering Cancer Center (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 12-353
Record Dates: First submitted 2012-11-04; First posted 2012-11-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Advanced; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating Tumor Cells (CTCs)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC: Subjects with advanced NSCLC, will undergo blood draw
  Interventions: Device: Circulating tumor cell chip

INTERVENTIONS:
Device: Circulating tumor cell chip — three tubes (6 teaspoons) of peripheral blood are drawn and are analyzed using the CTC chip
  Other Names: Herringbone circulating tumor cell chip, herringbone CTC chip, HBCTC chip

SUMMARY:
The purpose of this research study is to determine if the EGFR mutation can be detected in CTCs. CTCs are cancer cells that are shed from solid tumors and float freely in the bloodstream. A device called the CTC-chip has been developed to find CTCs in the blood of patients with cancer. This is an experimental device. Using this device, the investigators will test participants' blood to try and find CTCs with the EGFR mutation and compare them with the results from the biopsy your doctor has recommended. The long-term goal of this research is to develop a way to test for the EGFR mutation that is less invasive than a tumor biopsy.

DETAILED DESCRIPTION:
In order to participate in this study you need to have a diagnosis of NSCLC that has spread or is unable to be surgically removed. In addition, your cancer must have an EGFR mutation and you must have a scheduled (or recently performed) biopsy to check on the presence of any other mutations related to targeted drug resistance.

After you sign consent to participate in this study we will draw a blood sample (three tubes of blood). This is about 6 teaspoons of blood.

The number of CTCs in your blood will not be reported to you since it is not known if this number has any meaning or if it impacts your medical care in any way. These results will not become part of your medical record. They will be kept in a separate, secure location.

We will collect information from your medical records and store it in a research record that we create about you. The study team will use this information to compare details about your medical history with the results of the experiments done on your blood.

Genetic material (DNA) will be removed from the CTCs found in your blood. This genetic material will be stored at the Massachusetts General Hospital and studied along with samples from other participants on this research study. Your samples will not be labeled with your name or any information that identifies you. Your samples will have a study-specific code number on them. The code linking your name to the sample will be kept in a secure location, available only to the investigators of the study and select study team members.

After the blood draw we will follow your status every 6 months by reviewing your medical records.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC that is metastatic or unresectable
* Have agreed to undergo a clinically recommended invasive repeat tumor itssue biopsy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Receiving treatment for NSCLC at one of the participating cancer centers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with detectable EGFR mutations in their CTCs | 2 years
  Calculate the number of patients in the study population with detectable EGFR mutations in the CTCs in order to demonstrate the feasibility of testing for EGFR mutations from captured CTCs
Number of patients with CTC-derived EGFR genotyping matching their tumor-derived EGFR genotyping | 2 yearss
  Determine the concordance of EGFR genotyping from CTCs compared to tumor tissue

SECONDARY OUTCOMES:
Number of patients with EGFR gentoype results detectable from plasma cfDNA | 2 years
  Explore the feasibility of EGFR genotyping from plasma circulating free DNA (cfDNA)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas